CLINICAL TRIAL: NCT05484440
Title: Intervention Program With Perpetrators of Intimate Partner Violence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Minho (Other)
Responsible Party: Principal Investigator, Olga Cunha, Principal Investigator, University of Minho
Allocation: Non-Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: CE.CSH 102/2018
Record Dates: First submitted 2022-06-21; First posted 2022-08-02 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Intimate Partner Violence
Keywords: Intimate partner violence; Perpetrator; Intervention program

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group cognitive-behavioral intervention plus individual Motivational Interviewing (Experimental): Group participants will participate in six individual sessions based on Motivational Interviewing techniques (60 minutes each) and then in 18 group sessions based on psychoeducational and cognitive-behavioral techniques (90 to 120 minutes each). Groups will be composed of 6 to 10 participants. The intervention will be delivered weekly.
  Interventions: Other: Psychological
- Group cognitive-behavioral intervention (Experimental): Group participants will participate in 18 group sessions based on psychoeducational and cognitive-behavioral techniques (90 to 120 minutes each). Groups will be composed of 6 to 10 participants. The intervention will be delivered weekly.
  Interventions: Other: Psychological
- Treatment as usual (TAU) (No Intervention): Group participants will receive the usual treatment delivered by different institutions (e.g., correctional services, probation services, child protection services) as the participants of this study are justice-involved individuals (i.e., perpetrators of intimate partner violence).

INTERVENTIONS:
Other: Psychological
  Arms: Group cognitive-behavioral intervention; Group cognitive-behavioral intervention plus individual Motivational Interviewing

SUMMARY:
The current project aims to develop, implement and assess the effectiveness of an intervention program for perpetrators of intimate partner violence (both volunteers and court-mandated) that incorporates Motivational Interviewing techniques (MIT) as well as cognitive-behavioral and psychoeducational strategies implemented in a community setting. The intervention focuses on ending violence against the intimate partner and promoting the batterer's personal and social skills. The study uses pre- and post-treatment measures, with an experimental group (intervention) and two control groups (a group without intervention and a group without MIT). Data were collected at pre-test, post-test, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* being an adult male;
* having perpetrated physical, psychological, and/or sexual violence against a female intimate partner or ex-partner;
* be able to read and write.

Exclusion Criteria:

* psychotic disorders;
* cognitive impairment;
* psychological and/or personality disorders;
* substance abuse.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-01 (Actual); Primary Completion 2022-09 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Perpetration of abuse against intimate partner | 18 weeks
  Marital Violence Inventory (IVC) - Total scores range between 0 and 40. Higher scores mean a higher frequency of intimate partner violence.
Attitudes towards intimate partner violence | 18 weeks
  Attitudes towards Marital Violence Scale (ECVC) - Total score ranges between 25 and 125. Higher scores mean more supportive attitudes towards intimate partner violence.
Psychopathological symptoms | 18 weeks
  Bref Symptom Inventory (BSI) - BSI includes nine dimensions and three global indexes. Higher scores mean more psychopathological symptoms.
Coping skills | 18 weeks
  Coping scale - Total score ranges between 13 and 52. Higher scores mean better coping skills.
Risk of intimate partner violence | 18 weeks
  Spouse Abuse Risk Assessment (SARA) - Total scores range between 0 and 40. Higher scores mean a higher risk of intimate partner violence.
Motivation to change | 18 weeks
  University Rhode Island Change Assessment - Domestic Violence - Revised (URICA-DV-R) - URICA-DV-R includes a Readiness to Change Index - higher scores mean higher readiness to change.

SECONDARY OUTCOMES:
Self-esteem | 18 weeks
  Rosenberg Self-esteem scale (RSES) - Total scores range between 10 and 40. Higher scores mean higher self-esteem.
Self-concept | 18 weeks
  Self-concept inventory (ICAC) - Total scores range between 20 and 100. Higher scores mean higher self-concept.
Aggression | 18 weeks
  Buss-Perry Aggression Questionnaire (BPAQ) - Total scores range between 29 and 145. Higher scores mean higher levels of aggression.

CONTACTS AND LOCATIONS:
Locations (2):
- Portugal (2):
  - Associação de Psicologia da Universidade do Minho, Braga, None Selected
  - Junta de Freguesia Aver-o-Mar, Póvoa de Varzim

IPD SHARING:
Plan to Share IPD: No